CLINICAL TRIAL: NCT06669234
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of ALN-F1202, an siRNA Against Factor XII, in Healthy Adults
Brief Title: Phase 1 Safety and Tolerability Study of ALN-F1202 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-F1202-HV-2412; 2024-515286-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ALN-F1202 (Experimental): Randomized as described in the protocol Escalating Cohorts including Optional Cohorts
  Interventions: Drug: ALN-F1202
- Placebo (Experimental): Randomized as described in the protocol
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: ALN-F1202 — Administered per the protocol
  Arms: ALN-F1202
Drug: Matching Placebo — Administered per the protocol
  Arms: Placebo

SUMMARY:
This clinical research trial will evaluate the safety and tolerability of an experimental drug, ALN-F1202, in healthy participants.

The purpose of this trial is to learn about how safe and tolerable the experimental drug is. The trial is looking at several other research questions, including:

* What side effects may happen from taking the experimental drug?
* How much experimental drug is in the blood at different times?
* Whether the body makes antibodies against the experimental drug (which could make the drug less effective or could lead to side effects).
* What is the best dose of the experimental drug?

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a body mass index between 18 and 32 kg/m2, inclusive
2. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms (ECGs) performed at screening and/or prior to administration of initial dose of study drug
3. Is in good health based on laboratory safety testing obtained at the screening visit, as described in the protocol
4. Normal aPTT, normal PT, and normal platelet counts at screening period and at day -1 as defined by the local laboratory
5. Hemoglobin values at screening period and at day -1 as described in the protocol

Key Exclusion Criteria:

1. History of any major surgical procedure or clinically significant physical trauma, in the opinion of the investigator, that may pose a risk to the participant by study participation
2. Whole blood donation within the previous 56 days or plasma donation within the previous 7 days prior to screening
3. History of clinically significant bleeding, requiring hospitalization or blood products, that in the opinion of the investigator may pose a risk to the participant by study participation
4. History of bleeding diathesis as described in the protocol
5. Members of the clinical site study team and/or his/her immediate family, unless prior approval granted by the sponsor
6. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study

NOTE: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 190 Days
Severity of TEAEs | Up to 190 Days

SECONDARY OUTCOMES:
Change in activated Partial Thromboplastin Time (aPTT) | Baseline up to 190 Days
Change in Prothrombin Time (PT) | Baseline up to 190 Days
Concentration of combined ALN-F1202 and metabolites in plasma | Up to 190 Days
Extent of urinary excretion of combined ALN-F1202 and metabolites | Within 24 hours of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Center for Clinical Pharmacology University Hospitals Leuven (UZ Leuven), Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/